CLINICAL TRIAL: NCT03688035
Title: Prospective Study on the Potential of Circulating Tumor DNA to Assess the Tumor Response to Neoadjuvant Chemotherapy in Breast Cancer Patients
Brief Title: Potential of Circulating Tumor DNA to Assess the Tumor Response to Neoadjuvant Chemotherapy in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhiyong Yu (Other)
Responsible Party: Sponsor-Investigator, Zhiyong Yu, Director of the Breast Surgery Ⅰ, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Other Study IDs: ShandongCHI-08
Record Dates: First submitted 2018-08-30; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer; Neoadjuvant Chemotherapy; Circulating Tumor DNA
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — tissue samples from the surgery and blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is the most common malignant tumor in women worldwide,and there exist a large part of patients need to receive neoadjuvant chemotherapy(NAC) before the curative surgery.Circulating tumor DNA(ctDNA) is the circulating free DNA in the blood that originates from cancers,and it can be detected by modern technologies in plasma.In this prospective study,investigators aim to observe the correlation between tumor response to neoadjuvant chemotherapy and ctDNA.

DETAILED DESCRIPTION:
Women with node-positive breast cancer are at high risk for recurrence. Neoadjuvant chemotherapy is traditionally for locally advanced disease, converting an inoperable tumor to a resectable one.In the present study, investigators will focus on breast cancer patients whose primary tumors are large or have lymph node metastases and need to receive neoadjuvant chemotherapy from 2018 to 2019. Circulating tumor DNA(ctDNA) will be obtained from peripheral blood,and the blood samples will be taken before the neoadjuvant chemotherapy、during the chemotherapy、 before the surgery and post surgery visit (within 24 hours after surgery) .Investigators will collect tissue samples both from the breast lump biopsy and the curative surgery. Investigators aim to investigate whether circulating tumor DNA is a sensitive marker to monitor the efficacy of neoadjuvant chemotherapy in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing neoadjuvant chemotherapy
* Age: 18-70 yrs
* Any menopausal status
* Any hormone receptor status
* Invasive breast cancer proven histologically at diagnosis (before neoadjuvant chemotherapy):
* Locally advanced tumor
* Patients who received 6 to 8 cycles of neoadjuvant chemotherapy.

Exclusion Criteria:

* Failed to retain blood sample before NAC
* Lost more than 2 blood samples during NAC

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer patient receiving NAC in Shandong Cancer hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-09-20 (Estimated); Primary Completion 2019-09-20 (Estimated); Study Completion 2019-09-20 (Estimated)

PRIMARY OUTCOMES:
dynamic changes of plasma ctDNA mutant copies by a panel of 363 cancer-related genes | From patients recruited into the research until the surgury complete ,assessed up to 26 weeks.
  To assess the changes of ctDNA mutant copies during the process of our observation,and to find out the relationship between ctDNA and tumor response to neoadjuvant chemotherapy

SECONDARY OUTCOMES:
disease free survival after surgery | Up to 5 years
  To observe the duration from the end of curative surgery to local recurrence or distant metastasis of breast cancer. Patients were followed up every six months in first three years, then followed up once a year.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Yu, PHD, Study Chair — Shandong Cancer Hospital and Institute; Zhaoyun Liu, MD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China